CLINICAL TRIAL: NCT00382486
Title: Low Dose Ex-Vivo X-Irradiation of the Allograft and Simultaneous Bone Marrow Cell Infusion to Enhance Intestinal/Multivisceral Allograft Survival
Brief Title: Low Dose Irradiation for Small Bowel Transplant
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Other Study IDs: 0311041
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Irreversible Intestinal Failure; Allograft Rejection
Keywords: Intestinal transplant; Bone marrow; Irradiation of allograft

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Reduce the risk of allograft rejection

SUMMARY:
The specific aims of this study is to improve short and long-term patient and graft survival, to reduce the incidence and severity of allograft rejection, to reduce the incidence of infection and to reduce and/or eventually eliminate the need for long-term immunosuppression.

DETAILED DESCRIPTION:
The rationale behind this study involves the need to better manage rejection in the intestinal allograft recipient. Although tacrolimus based immunosuppression has made intestinal transplantation feasible, the requisite need for chronic high dose immunosuppression in order to control rejection has inhibited the wide spread clinical use and practicality of intestinal/multivisceral transplantation. The measures needed to prevent graft loss have frequently resulted in lethal infections, the leading cause of death. This trial is significant for determining if this new strategy of allograft immune-modulation with low dose ex-vivo irradiation and simultaneous done bone marrow cell infusion will favorably affect short and long term outcomes by reducing the risk of allograft rejection.

This trial is offered to all patients with irreversible intestinal failure who must undergo intestinal, combined liver-intestinal, and multivisceral transplantation at the University of Pittsburgh Medical Center. Patients are recruited through the referral system and no cold calling is carried out. Patient confidentiality is maintained by the use of codes to identify the study participants. All data is stored in a locked filing cabinets as a means to protect participants against a breach of confidentiality. This trial involves ex-vivo low dose irradiation of the intestinal allograft with or without adjunct donor bone marrow cell infusion. An intravenous bone marrow cell infusion is prepared form the thoracolumbar vertebral bodies harvested from cadaveric donors. Control subjects will be those who refuse to be enrolled in the study or those for whom donor bone marrow is not available. All patients will be treated perioperatively with thymoglobulin, a rabbit polyclonal anti-lymphocyte globulin at a dose of 5-10 mg/kg. Tacrolimus will be given in a standard fashion and from the outset as a single monotherapeutic agent to prevent early allograft rejection and promote graft acceptance. All patients will be monitored for rejection, graft function, opportunistic infections and GVHD. Surveillance endoscopy with guided mucosal biopsies will be obtained according to the standard protocol. Attention will be paid for any clinicopathologic changes suggestive of acute or chronic irradiation injuries.

The study closed for enrollment as of 9/30/03.

ELIGIBILITY:
Inclusion Criteria:

* all patients between 17 and 70 who are diagnosed with intestinal failure awaiting intestinal/multivisceral transplant

Exclusion Criteria:

* active systemic/abdominal infections
* incurable malignancy
* acquired immune deficiency syndrome
* severe cardiopulmonary insufficiency
* current alcoholism
* pregnant female

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2001-07; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kareem M Abu-Elmagd, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States